CLINICAL TRIAL: NCT00756236
Title: A Comparison of the Effect of Intraoperative Administration of Metoprolol or Esmolol on General Anesthetic Requirement
Brief Title: A Comparison of the Effects of Intraoperative Administration of Metoprolol or Esmolol on General Anesthetic Requirement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 1638
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-06

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia | interventions — Metoprolol; esmolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- M-Group (Experimental): Patients were randomly assigned to Metoprolol Group. The drug was dispensed in 60ml & 5ml syringes of 0.9% NaCl and 1mg/ml Metoprolol. Investigators and patients were blinded to the group assignment.
  Interventions: Drug: Metoprolol
- E-Group (Experimental): Patients were randomly assigned to Esmolol Group. The drug was dispensed in 60ml & 5ml syringes of 0.9% NaCl and 10mg/ml Esmolol. Investigators and patients were blinded to the group assignment.
  Interventions: Drug: Esmolol
- P-Group (Placebo Comparator): Patients were randomly assigned to this group. Patients received 0.9% NaCl only. To maintain the blind, 0.9% NaCl was also dispensed in 60ml & 5ml syringes.
  Interventions: Drug: P-Group

INTERVENTIONS:
Drug: Metoprolol — 60ml syringes of 0.9% NaCl, 5ml syringes of metoprolol at 1mg/ml concentration
  Other Names: M-Group
  Arms: M-Group
Drug: Esmolol — 60ml syringes of esmolol at 10 mg/ml concentration, 5ml syringes of 0.9% of NaCl
  Other Names: E-Group
  Arms: E-Group
Drug: P-Group — 0.9%NaCl dispensed in 60ml & 5ml syringes
  Other Names: Placebo Comparator
  Arms: P-Group

SUMMARY:
We will compare three study groups receiving metoprolol, esmolol, or placebo. Level of anesthesia will be titrated to achieve the same range of BIS value in all groups. Our hypothesis is that the metoprolol and esmolol groups will require a lower level of anesthetic agent to achieve the targeted BIS range, compared to the placebo group.

Our objective is to clarify if metoprolol, in a dose range used for perioperative cardiac protection, decreases anesthetic requirement.

DETAILED DESCRIPTION:
Beta-receptor antagonists are commonly used in the perioperative setting. These agents have been shown to decrease the incidence of perioperative myocardial ischemia and are recommended by a recent practice guideline in certain patient groups.1 Besides protection from ischemia, there are other situations where beta-receptor antagonists are used intraoperatively such as control of the sympathetic response to tracheal intubation and certain types of surgical stimuli.

There is new evidence suggesting that administration of esmolol, a short-acting beta-receptor antagonist, might reduce the actual anesthetic requirement. This was initially shown by studies in which esmolol decreased the amount of anesthetic required to prevent movement after skin incision.2;3 Subsequent studies used bispectral index (BIS) as an endpoint and demonstrated decreased BIS values in subjects receiving esmolol during general anesthesia. 4;5

This anesthetic-sparing effect observed with esmolol has not been prospectively studied with other beta-receptor antagonists. Since perioperative beta-blockade is commonly achieved using longer acting agents such as metoprolol or atenolol, it is clinically relevant to understand the effects of these medications on anesthetic requirement. We aim to conduct a prospective, randomized, controlled, double-blind study to compare the anesthetic-sparing effect of metoprolol and esmolol administered intraoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Being older than 18 but, not older than 75
* Scheduled for surgery under general anesthesia
* Duration of surgery scheduled as 2 hours or longer

Exclusion Criteria:

* Intracranial or intrathoracic surgery (due to difficulty using a BIS monitor or frequent need for beta-receptor antagonism)
* Indication for perioperative beta-receptor antagonism
* Current use of calcium-channel antagonists
* History of coronary artery disease
* History of reactive airway disease
* History of diabetes or other disorders of glucose metabolism
* Reported allergy to any of the study drugs
* Reported substance abuse (except nicotine and caffeine)
* Use of monoamine oxidase (MAO) inhibitor drugs
* Hypersensitivity to metoprolol, esmolol and related derivatives, or to any of the excipients of either.
* Hypersensitivity to other beta-blockers (cross-sensitivity between beta-blockers can occur).
* Sick-sinus Syndrome.
* Heart block greater than first degree, cardiogenic shock, and overt cardiac failure.
* Significant first-degree heart block (P-R interval greater than or equal to 0.24 sec; systolic pressure < 100mmHg; or moderate- to-severe cardiac failure).
* Severe peripheral arterial circulatory disorders.
* Pheochromocytoma.
* Baseline heart rate of < 60
* Systolic pressure less than 100 mm Hg
* Pregnant women
* Prisoners

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-10; Primary Completion 2015-09-02 (Actual); Study Completion 2015-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pramod Chetty, MD, Principal Investigator — Faculty, Anesthesiology
Locations (1):
- Univeristy of Oklahoma Health Sciences Center Dept. Anesthesiology, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of Oklahoma Health Sciences Center — http://www.ouhsc.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were consented at the pre-surgical clinical visit if they were outpatients. Inpatients were consented while they were in the hospital. Each patient were provided with a copy of the informed consent and be given at least 12 hours to make a decision.
Pre-assignment Details: Group assignments were randomized by a pharmacist who also prepared the study drugs. Investigators and subjects were blinded to the group assignment.
Period: Overall Study
Arm/Group | M-Group | E-Group | P-Group
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | M-Group | E-Group | P-Group | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 18 | 17 | 55
  >=65 years | 0 | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 44 (13.3) | 49 (11.8) | 48 (15.2) | 46.8 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 14 | 43
  Male | 8 | 3 | 6 | 17
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve of etSEV Over the First Hour
Description: We will measure the amount of Sevoflurane used to achieve the same level Bispectral Index. Each patient will have their percentage of sevoflurane in expired breath measured every 5 minutes for 2 hours, resulting in 24 data points per person. The primary endpoint will be area under the curve (AUC) for each subject for the first hour.
Time Frame: Every 5 minutes for 2 hours
Measure: Mean (Standard Deviation); unit: percent*hour
Arm/Group | M-Group | E-Group | P-Group
Number analyzed (Participants) | 20 | 20 | 19
percent*hour | 1.77 (0.38) | 1.46 (0.29) | 1.73 (0.47)

ADVERSE EVENTS:
Time Frame: From start of the surgical procedure to one day after the surgery.
Description: Inpatients will be seen the day after the surgical procedure to assess signs of adverse effects. Range of heart rate and blood pressure since the operation will be recorded. Patients will be asked about any incidence of wheezing since the surgery. Patients' chest will be auscultated at this visit to detect wheezing.
Arm/Group | M-Group | E-Group | P-Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
1. Surgical stimulus was not standardized.
2. ß-blockade in Group M was not as uniform as that of Group E.
3. There was considerable variation in achieving the target BIS level.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No